CLINICAL TRIAL: NCT07053124
Title: Diagnostic Efficiency Comparation of Hand-Drawn Navigation and Virtual Navigation for Peripheral Pulmonary Nodules: A Prospective, Randomized, Parallel-Controlled, Global Multicenter Clinical Study
Brief Title: Diagnostic Efficiency Comparasion of Hand-Drawn Navigation and Virtual Navigation for Peripheral Pulmonary Nodules
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, Professor, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Hand-drawn navigation
Record Dates: First submitted 2025-06-17; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Pulmonary Nodules
Keywords: Peripheral pulmonary nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand-drawn group (Experimental): Hand-drawn navigation was employed for diagnosing patients with PPN .
  Interventions: Other: Hand-drawn navigation
- VBN group (Active Comparator): Virtual bronchosocopy navigation was employed for diagnosing patients with PPN .
  Interventions: Other: Virtual bronchoscopy navigation

INTERVENTIONS:
Other: Hand-drawn navigation — Hand-drawn navigation employed for diagnosing patients with PPN in Hand-drawn group.
  Arms: Hand-drawn group
Other: Virtual bronchoscopy navigation — Virtual bronchoscopy navigation employed for diagnosing patients with PPN in VBN group.
  Arms: VBN group

SUMMARY:
Peripheral pulmonary lesions (PPLs) refer to isolated or localized lesions located in the outer one-third of the lung field. Their qualitative diagnosis is a key link in the early screening and precise treatment of lung cancer. However, due to the deep location, small size (especially those with diameters < 2 cm), and unclear relationship with bronchi of peripheral pulmonary lesions, traditional bronchoscopy is difficult to directly reach the lesion, resulting in a relatively low positive rate of biopsy. Moreover, although conventional imaging examinations (such as CT) can locate the lesions, they cannot provide a histological diagnostic basis. Percutaneous puncture under CT guidance has high risks such as pneumothorax, bleeding and pleural reaction, and has low efficiency in locating multiple lesions.

At present, there are various auxiliary techniques for the diagnosis of peripheral pulmonary nodules, each with its own advantages and disadvantages:

1. Image-guided techniques: Although traditional CT-guided percutaneous biopsy is intuitive in terms of localization, it has high complication risks and limited applicability for nodules close to the mediastinum or blood vessels.
2. Radial Bronchial Endobronchial Ultrasound (RP-EBUS): Combined with a guide sheath (GS), it can increase the positive rate of peripheral nodule biopsy (the weighted diagnostic rate without fluoroscopy can reach 70%), but it relies on the operator's familiarity with bronchial anatomy and is difficult to solve complex bronchial path planning problems alone.
3. Virtual Bronchoscopy Navigation (VBN): VBN generates virtual bronchial paths based on CT three-dimensional reconstruction, significantly shortening the operation time and improving the diagnostic rate (62.5%-84.4%, overall 73.8%). However, its limitations are obvious: it relies on high-quality CT images and is sensitive to respiratory motion artifacts; it cannot be adjusted in real time, and during the operation, it is prone to deviate from the navigation map due to anatomical variations or secretions, with high equipment costs and difficulty in popularization in grassroots hospitals.
4. Electromagnetic Navigation Bronchoscopy (ENB): ENB achieves precise navigation through electromagnetic positioning, with a diagnostic rate of up to 70%-80%, but the equipment is expensive (single consumable cost is about 1-20,000 yuan), and it needs to be combined with intraoperative fluoroscopy.
5. Robotic-assisted bronchoscopy navigation: Emerging technologies such as robotic-assisted navigation offer good stability and high precision in control, but they are complex in terms of technology and expensive in terms of equipment. Currently, they are only available in large medical centers in China.

Hand-drawn Mapping Navigation is a manual drawing technique based on preoperative CT images. By marking the directions of bronchial branches and the positions of nodules, it provides the surgeons with intuitive path planning. Studies have shown that hand-drawn navigation combined with RP-EBUS can shorten the time for bronchoscopy to reach the biopsy site from 8.89 ± 4.09 minutes to 6.32 ± 3.10 minutes (P < 0.001), and bronchial grading and hand-drawn navigation are independent influencing factors. Compared with VBN, its advantages lie in: low cost, only requiring pen and paper or electronic drawing tools, high flexibility, and the ability to adjust the path in real time in combination with the surgeon's experience; no reliance on complex software or hardware equipment, suitable for areas with limited resources. Currently, there have been many studies exploring the clinical value of hand-drawn mapping navigation maps and comparing them with VBN. However, most of the existing studies are limited to single-center retrospective analyses and lack prospective control evidence compared with VBN.

This study aims to compare the clinical application value of hand-drawn navigation and VBN in the diagnosis of peripheral pulmonary nodules through a randomized controlled trial. The main objective is to evaluate the differences in clinical application between the hand-drawn navigation group and the VBN group in terms of bronchoscopy arrival time, positive biopsy rate, and complication occurrence rate; analyze the applicability of the two techniques in different bronchial grade nodules, etc. The study results will provide evidence-based basis for optimizing the diagnosis and treatment pathway of peripheral pulmonary nodules and lay a foundation for the development of low-cost precise navigation technology.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years;
2. Patients with pulmonary nodule and nodule size >8mm but ≤ 30mm, bronchus level of the nodule ≥ grade 5, who are scheduled to undergo bronchoscopy biopsy for definitive diagnosis;
3. In the judgment of investigator that the nodule is difficult to reach with conventional bronchoscopy and bronchoscopy guidance technology is needed.

Exclusion Criteria:

1. Contraindications for bronchoscopy examination;
2. Other situations what investigators consider inappropriate for participation.1.Contraindications for bronchoscopy examination; Other situations what investigators consider inappropriate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Intermediate Diagnosis yield | 6 monthes after procedure
  Intermediate Diagnosis yield, which is calculated based on the follow-up data of cases where NSB was detected by bronchoscopy only. Only cases where subsequent biopsy or imaging examination confirmed non-malignant diagnosis (NSBTN) will be classified as true negatives; cases without a clear diagnosis due to lack of follow-up will be regarded as non-diagnosed. Patients who fail to navigate but switch paths to continue the biopsy to achieve a diagnosis will not be counted as successful cases. The calculation formula is (TP + SPB + NSBTN) divided by the total number of procedures. The differences between the two groups will be compared

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhong CH, Su ZQ, Luo WZ, Rao WY, Feng JX, Tang CL, Chen Y, Chen XB, Fan MY, Li SY. Hierarchical clock-scale hand-drawn mapping as a simple method for bronchoscopic navigation in peripheral pulmonary nodule. Respir Res. 2022 Sep 14;23(1):245. doi: 10.1186/s12931-022-02160-0. PMID 36104691